CLINICAL TRIAL: NCT03691376
Title: A Phase I, Open Label Study Evaluating the Safety and Efficacy of Adoptive Transfer of Autologous NY-ESO-1 CD8-TCR Engineered T Cells and NY-ESO-1 CD4-TCR Engineered Hematopoietic Stem Cells (HSC) After a Myeloablative Conditioning Regimen, With Administration of IL-2 in Patients With Recurrent or Treatment Refractory Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Genetically Engineered Cells (NY-ESO-1 TCR Engineered T Cells and HSCs) After Melphalan Conditioning Regimen in Treating Patients With Recurrent or Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i 287616; NCI-2018-01758 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 287616 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Platinum-Sensitive Fallopian Tube Carcinoma; Platinum-Sensitive Ovarian Carcinoma; Platinum-Sensitive Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Refractory Fallopian Tube Carcinoma; Refractory Ovarian Carcinoma; Refractory Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — aldesleukin; Cell- and Tissue-Based Therapy; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (autologous NY-ESO-1 engineered T and HSC) (Experimental): Patients receive melphalan IV over 30 minutes on day -1. Patients then receive autologous NY-ESO-1 CD4-TCR CD34+ HSC IV on day 0 and autologous NY-ESO-1-specific CD8-positive T lymphocytes IV between days 7 and 21. Patients also receive aldesleukin SC BID for 14 days on the following day after the T cell infusion (between days 8 and 22).
  Interventions: Biological: Aldesleukin; Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes; Other: Cellular Therapy; Drug: Melphalan

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; recombinant human interleukin-2
Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes — Given IV
Other: Cellular Therapy — Given autologous NY-ESO-1 CD4-TCR CD34+ HSC IV
  Other Names: Cell Therapy
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813

SUMMARY:
This phase I trial studies the best dose and side effects of NY-ESO-1 T cell receptor (TCR) engineered T cells and how well they work with NY-ESO-1 TCR engineered hematopoietic stem cells (HSCs) after melphalan conditioning regimen in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back (recurrent) or does not respond to treatment (refractory). The melphalan conditioning chemotherapy makes room in the patient's bone marrow for new blood cells and blood-forming cells (stem cells) to grow. Giving NY-ESO-1 TCR T cells and stem cells after the conditioning chemotherapy is intended to replace the immune system with new immune cells that have been redirected to attack and kill the cancer cells and thereby improve immune system function against cancer. Giving NY-ESO-1 TCR engineered T cells and HSCs after melphalan may work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of intravenous infusion of autologous peripheral blood mononuclear cells (PBMC) and CD34+ peripheral blood stem cells (PBSC) that have been genetically modified ex vivo to express NY-ESO-1 TCR, following a myeloablative conditioning regimen.

Ia. Assessment of toxicities using Common Toxicity Criteria (CTC) and definition of a maximum tolerated dose (MTD).

SECONDARY OBJECTIVES:

I. TCR engineered hematopoietic stem cell (HSC) engraftment. II. Functional assays for TCR transgenic cells. III. Progression-free survival (PFS) (compare with the duration of the PFS in the last treatment regimen).

IV. Durable tumor response in at least 30% of the patients defined as immune-related complete response (irCR) or immune-related partial response (irPR) by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) criteria at 6 months.

V. Long-term persistence of TCR transgenic cells (regardless of cell origin) as evidenced by > 5% of CD3 lymphocytes being NY-ESO-1 specific by major histocompatibility complex (MHC) tetramer assay at 3 and 6 months.

VI. Discrimination of TCR transgenic cells resulting from retrovirally-transduced mature lymphocytes and lentivirally-transduced HSCs and their phenotyping.

VII. Long term monitoring for replication competent retrovirus and lentivirus. VIII. Analysis of viral insertion sites in long term persisting NY-ESO-1 TCR clones: absence of a clonal expansion of TCR transgenic cells with a particular transgene insertion site (defined as a clone comprising > 20% of all PBSC-derived gene-marked cells).

IX. Gut microbiota pre and post treatment to evaluate the role of microbiota on the therapeutic efficacy of the proposed therapy.

OUTLINE: This is a dose-escalation study of autologous NY-ESO-1-specific CD8-positive T lymphocytes.

Patients receive melphalan intravenously (IV) over 30 minutes on day -1. Patients then receive autologous NY-ESO-1 CD4-TCR CD34+ HSC IV on day 0 and autologous NY-ESO-1-specific CD8-positive T lymphocytes IV between days 7 and 21. Patients also receive aldesleukin subcutaneously (SC) twice daily (BID) for 14 days on the following day after the T cell infusion (between days 8 and 22).

After completion of study treatment, patients are followed up every 6 months for 5 years, then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of platinum-sensitive or platinum-resistant recurrent or refractory epithelial ovarian, primary peritoneal or fallopian tube carcinoma and have progressed, relapsed, or recurred through at least one or more prior lines of standard-of-care therapies. For platinum sensitive patients, the standard of care therapies include additional platinum-containing regimens and bevacizumab
* Have been informed of other treatment options
* Must be HLA- A*02.1 and HLA-DP*04 positive. Retesting is not required for patients who have previous documented positivity
* Patient's tumor must be positive by histological or molecular assay for NY-ESO-1
* Have an Eastern Cooperative Oncology group (ECOG) performance status of 0 or 1
* Life expectancy of > 4 months
* At least 4 weeks from prior chemotherapy, radiotherapy or immunotherapy, or prior investigational agents
* Must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Must have adequate venous access for apheresis (pheresis catheter placement for cell collection is allowed)
* Since the study drug may affect pregnancy since it targets proteins present during development, women of childbearing potential are requested to use acceptable methods of birth control for the duration of the study and until persistence of the study drug is no longer detected in the patient by polymerase chain reaction (PCR). This may be a period of several years. Methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception. It is recommended that a combination of two methods be used
* Leukocytes >= 3 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 2 x upper limit of normal (ULN); if creatinine level > 2 x ULN, then creatinine clearance must be > 60 mL/min
* Patient must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participant must agree to and arrange for a caregiver (age >= 18 years old) available 24 hours a day/ 7 days a week and arrange for lodging within 45 minutes drive to Roswell Park and transportation for a period of time after discharge from the hospital. The exact amount of time will depend on the individual status as determined by the treating physician

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Known cases of clinically active brain metastases (brain magnetic resonance imaging [MRI] as clinically indicated). Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study
* Prior malignancy (except non melanoma skin cancer) within 3 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin 2, interferon alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study entry

  * NOTE: Recent or current use of inhaled steroids and topical steroids are not exclusionary. If subjects are prescribed a brief course of oral corticosteroids, the use should be limited to less than 7 days. Use of steroids before apheresis and immune assessment blood draws should be discouraged as it will affect white blood cell function
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV) as defined below, due to the immunosuppressive effects of chemo-conditioning used and the unknown risks associated with viral replication

  * Positive serology for HIV
  * Active hepatitis B infection as determined by test for hepatitis B surface antigen (Ag)
  * Active hepatitis C. Patients will be screened for HCV antibody. If the HCV antibody is positive, a screening HCV ribonucleic acid (RNA) by any reverse transcriptase (RT) PCR or branched deoxyribonucleic acid (bDNA) assay must be performed at screening by a local laboratory with a Clinical Laboratory Improvement Act (CLIA) certification or its equivalent. Eligibility will be determined based on a negative screening value. The test is not required if documentation of a negative result of a HCV RNA test performed within 60 days prior to screening is provided.
  * Serology (CMV IgG) positive for active CMV
* Received any previous gene therapy using an integrating vector within 6 months
* Pregnancy or breast-feeding
* Lack of availability of a patient for immunological and clinical follow up assessment
* Evidence or history of significant cardiac disease (including myocardial infarction [MI] in the past 6 months, significant cardiac arrhythmia, stage III or IV congestive heart failure [CHF]). Cardiac stress test will be done if clinically indicated. (The specific test to be chosen at the discretion of the principal investigator [PI])
* Patients with pulmonary function test abnormalities as evidenced by a forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) < 70% of predicted for normality will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 9 months post infusion
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles.
Maximum tolerated dose (MTD) | Up to 9 months post-infusion
  Dose limiting toxicities will be used in the estimation of the MTD and the accompanying of the dose escalation decisions. The frequency of toxicities will also be tabulated for the dose estimated to be the MTD.

SECONDARY OUTCOMES:
Change in Immunological parameters associated with T cell persistence | Baseline up to 15 years
Tumor response rates to treatment | Up to 15 years
  Based on the immune-related Response Evaluation Criteria in Solid Tumors criteria.
Progression-free survival | From start of the treatment until the first occurrence of confirmed progression, assessed up to 15 years
  Will calculate the median progression free survival and the corresponding 95% confidence interval.
Overall survival | From start of the treatment until death, assessed up to 15 years
Duration of response | Up to 15 years
Appearance of target antigen/major histocompatibility complex loss variants upon disease recurrence | Up to 15 years
  NY-ESO-1 expression will be evaluated by quantitative reverse transcriptase polymerase chain reaction (Q-RT-PCR) and/or immunohistochemistry. HLA-A*0201 and -DP*04 expression on samples will be evaluated by immunohistochemistry.
Assessment of bioactivity | Baseline up to 15 years
  measure pre and post treatment percentage of selective migration into the tumor sites
Assessment of Immunological parameters associated with functionality | Baseline up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States